CLINICAL TRIAL: NCT01552655
Title: Breast Cancer Recurrence - the Accuracy of Dual-time PET/CT
Acronym: BREAC-AUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Kirsten Falch, Medical Technologist, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: BREAC-AUT
Record Dates: First submitted 2012-02-28; First posted 2012-03-13 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Breast Cancer Recurrent
Keywords: Dual-time PET/CT; Breast cancer recurrence; Bone scintigraphy; CT thorax upper abdomen

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dual-time PET/CT (Other)
  Interventions: Radiation: Dual-time PET/CT (low-dose)

INTERVENTIONS:
Radiation: Dual-time PET/CT (low-dose) — 4 MBq/kg 18F-flour-deoxyglucose administered iv. PET/CT-scans performed 60 min and 180 min after injection.

SUMMARY:
The purpose of this study is to elucidate the value of dual-time-point PET/CT in the recurrence of breast cancer and to determine whether the method is better than the modalities used in the standard work up.

150 patients with suspected breast cancer recurrence will be included. All patients will undergo dual-time-point PET/CT, CT of thorax and upper abdomen and bone scintigraphy. After completion of the examinations the early and the late PET/CT scan will be compared with each other, the diagnostic CT-scan and the bone scintigraphy. A verification of suspicious findings will be done by biopsy, if the area is accessible. If a biopsy cannot be obtained, the presence of recurrence will be verified with additional imaging follow-up to ensure the highest possible confidence. Sensitivity, specificity, accuracy, negative and positive predictive value (NPV/PPV) will be calculated for each modality (incl. early and late PET/CT).

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspected recurrence of breast cancer
* Blood glucose level less than 8,0 mmol/L

Exclusion Criteria:

* Disqualified patients
* Other malignancies
* < 18 years
* < 50 kg
* > 90 kg
* Pregnant or lactating
* Patients with permanent address outside of the Region of Southern Denmark
* Estimated inability to collaborate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic value of dual-time point 18FDG PET/CT in recurrent breast cancer | 2 years
  The sensitivity and specificity of dual-time point 18FDG PET/CT will be compared to conventional imaging modalities usually used in the work up of patients with suspected recurrent breast cancer. In this case CT of thorax and upper abdomen and bone scintigraphy.

SECONDARY OUTCOMES:
Diagnostic value of early and late 18FDG PET/CT respectively in recurrent breast cancer | 2 years
  The sensitivity and specificity of early (60 min post injection) and late (180 min post injection) 18FDG PET/CT respectively in patients with suspected recurrent breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Malene Hildebrandt, M.D., Principal Investigator — Dept. Nuclear Medicine, Odense University Hospital
Locations (1):
- Department of Nuclear Medicine, Odense University Hospital, Odense, Funen, Denmark

REFERENCES:
- [Derived] Vogsen M, Geneser S, Rasmussen ML, Horder M, Hildebrandt MG. Learning from patient involvement in a clinical study analyzing PET/CT in women with advanced breast cancer. Res Involv Engagem. 2020 Jan 6;6:1. doi: 10.1186/s40900-019-0174-y. eCollection 2020. PMID 31921443
- [Derived] Baun C, Falch K, Gerke O, Hansen J, Nguyen T, Alavi A, Hoilund-Carlsen PF, Hildebrandt MG. Quantification of FDG-PET/CT with delayed imaging in patients with newly diagnosed recurrent breast cancer. BMC Med Imaging. 2018 May 9;18(1):11. doi: 10.1186/s12880-018-0254-8. PMID 29743027